CLINICAL TRIAL: NCT00595153
Title: Determining Mechanisms of Asthma Through Detailed Analysis of Airway Secretions and Tissues
Brief Title: Study of the Mechanisms of Asthma
Acronym: MAST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UCSF CHR# H6788-30617
Record Dates: First submitted 2008-01-02; First posted 2008-01-16 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- B (Active Comparator): Asthmatics not on inhaled corticosteroids who will be put on an inhaled steroid during the study
  Interventions: Drug: Pulmicort
- A (No Intervention): Healthy, non-asthmatics who will not be put on any intervention
- C (Active Comparator): Asthmatics, who are already on inhaled corticosteroids who will be put on standardized dose of inhaled corticosteroids
  Interventions: Drug: Pulmicort

INTERVENTIONS:
Drug: Pulmicort — inhaled powder of inhaled corticosteroid, 1 puff (180mcg) twice a day for 8-10 weeks
  Other Names: Budesonide
  Arms: B; C

SUMMARY:
The purpose of this study is to identify the causes of asthma that were not previously suspected, to better understand the effects of inhaled steroids on asthma and to identify new way to treat asthma. In order to take advantage of the most current scientific expertise, we (scientists at UCSF) plan to work together with Genentech Inc. We believe that working with Genentech will provide the best chance of developing new treatments for asthma.

DETAILED DESCRIPTION:
Asthma is a common airway disease with persistent unmet needs on terms of treatment. Although many asthmatics enjoy good control of their disease by using regularly scheduled corticosteroid treatment, a significant minority do not achieve optimal control with steroids and suffer asthma exacerbations which can be severe and even fatal. Asthma pathophysiology is complex and involves multiple cell types and multiple signaling mechanisms. One approach to this complexity has been to study responses of isolated airway cells to experimental conditions which model asthmatic inflammation; another has been genetic manipulations of candidate mediators of asthma in inbred mice. These studies have yielded important insights about possible mechanisms of asthma in humans, but the relevance of these mechanisms to human disease has not always been proven, and it is possible that unsuspected mechanism have not yet been revealed by these approaches. In the studies proposed here we will take an experimental approach which takes advantage of the distinct clinical phenotype of human asthma, the ability to measure steroid response in asthma, the relative ease of collecting airway cells and tissues by bronchoscopy, and the availability of new technologies such as high density microarrays which have probes for all genes in the genome or proteomics which can identify all proteins present in a biologic sample. Using this approach, we will identify differential expression of genes and proteins in airway cells and tissues in asthma that can then be explored further in cell and animal model systems to determine their potential as drug targets in asthma. We further believe that our approach will identify previously unsuspected mechanisms of action of corticosteroids in airway cells and tissues in asthma. Presently, relatively little is known about why some asthmatics respond well and some poorly to steroids and closing this gap in knowledge will help identify candidate genes and proteins to target in order to address unmet therapeutic needs in asthmatics with steroid resistant asthma.

ELIGIBILITY:
Inclusion Criteria:

Group C:

* Male and female subjects between the ages of 18 and 70 years
* History of asthma
* Continuous treatment with inhaled corticosteroids for at least the 6-week
* Hyperreactivity to methacholine (provocative concentration of methacholine causing a 20% drop in forced expiratory volume in 1 second (PC20 FEV1) Methacholine ≤ 16.0 mg/mL).

Exclusion Criteria:

* History of asthma
* No use of oral or inhaled corticosteroids for the treatment of asthma in the past 6 weeks
* Hyperreactivity to methacholine (PC20 FEV1 Methacholine ≤ 8.0 mg/mL).
* At least one of the following symptoms, beta agonist use, or FEV1 criteria:

  * Asthma symptoms on at least two days per week; OR
  * Beta agonist use on at least two days per week; OR
  * Forced expiratory volume in 1 second (FEV1) < 85% predicted
* Subjects must be non-smokers (patients who have never smoked or patients who have not smoked for 1 year and have a total pack-year smoking history < 15 packs).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2007-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John V Fahy, M.D., M.Sc., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Solberg OD, Ostrin EJ, Love MI, Peng JC, Bhakta NR, Hou L, Nguyen C, Solon M, Nguyen C, Barczak AJ, Zlock LT, Blagev DP, Finkbeiner WE, Ansel KM, Arron JR, Erle DJ, Woodruff PG. Airway epithelial miRNA expression is altered in asthma. Am J Respir Crit Care Med. 2012 Nov 15;186(10):965-74. doi: 10.1164/rccm.201201-0027OC. Epub 2012 Sep 6. PMID 22955319
- See also: Airway Clinical Research Center website — http://airway.ucsf.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The MAST study enrolled 103 adults with asthma and 24 healthy controls between 8/2007 to 6/2011. Participants were seen in a clinical research center.
Pre-assignment Details: Steroid naïve asthmatics had bronchoscopy before and after an 8 week treatment with inhaled corticosteroids, and asthmatics already taking an inhaled corticosteroid had their treatment standardized for 8 weeks followed by a bronchoscopy. Healthy control subjects participated in a cross-sectional study for characterization and bronchoscopy.
Groups:
- Healthy Control: Healthy, non-asthmatics who will not be put on any intervention
- Steroid Naive Asthmatics: Asthmatics not on inhaled corticosteroids who will be put on an inhaled steroid during the study
  Pulmicort : inhaled powder of inhaled corticosteroid, 1 puff (180mcg) twice a day for 8-10 weeks
- Asthmatics on ICS Treatment: Asthmatics, who are already on inhaled corticosteroids who will be put on standardized dose of inhaled corticosteroids
  Pulmicort : inhaled powder of inhaled corticosteroid, 1 puff (180mcg) twice a day for 8-10 weeks
Period: Overall Study
Arm/Group | Healthy Control | Steroid Naive Asthmatics | Asthmatics on ICS Treatment
Started | 24 | 42 | 61
Completed | 20 | 26 | 36
Not Completed | 4 | 16 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Steroid Naive Asthmatics | Asthmatics on ICS Treatment | Total
Number analyzed (Participants) | 24 | 42 | 61 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 42 | 61 | 127
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (9.0) | 32.0 (11.6) | 39.0 (11.9) | 35.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 27 | 34 | 71
  Male | 14 | 15 | 27 | 56
Region of Enrollment [Number; unit: participants]
  United States | 24 | 42 | 61 | 127

OUTCOME MEASURES:

1. Primary Outcome: Gene Expression in Airway Secretions and Tissues
Description: The primary outcome measure for this study is the scaled mean value of three gene expression markers of IL-13 in the airway: PERIOSTIN, calcium-activated chloride channel regulator 1 (CLCA1), and plasminogen activator inhibitor-2 (SERPINB2). First, for each of the three interleukin-13 (IL-13) signature genes, the log (base-2) transformed relative expression value for each subject is measured using real-time polymerase chair reaction (PCR) and normalized with the geometric mean of 5 housekeeping genes. Next, these values are centered (by subtracting the mean for that gene) and scaled (by dividing by the standard deviation for that gene) so that each gene makes an equal, assay-independent contribution to the Th2 phenotype. Then, for each subject, the arithmetic mean of the three centered & scaled genes is calculated, producing the "three-gene-mean" metric.
Time Frame: Healthy Control: Visit 2 (at 1 week); Steroid Naive Asthmatics: Visit 2 (at 1 week); Steroid Treated Asthmatics: Visit 5 (at 9 weeks)
Population: Participants who met inclusion/exclusion requirements and completed all study activities were included in the analysis. Specifically, this included:
  1. Having a bronchoscopy with complete PCR on RNA from epithelial brush samples.
Measure: Mean (Standard Deviation); unit: Relative gene expression level
Arm/Group | Healthy Control | Steroid Naive Asthmatics | Asthmatics on ICS Treatment
Number analyzed (Participants) | 19 | 24 | 21
Relative gene expression level | -0.66 (0.36) | 0.54 (0.87) | -0.30 (0.60)

ADVERSE EVENTS:
Arm/Group | Healthy Control | Steroid Naive Asthmatics | Asthmatics on ICS Treatment
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/42 | 0/61
Other Adverse Events (participants affected / at risk) | 6/24 | 5/42 | 15/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Healthy Control (N=24) | Steroid Naive Asthmatics (N=42) | Asthmatics on ICS Treatment (N=61)
Increased asthma symptoms following medication hold (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0 (0) | 5 (60)
Did not tolerate switch of asthma controller medication (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0 (0) | 5 (60)
Respiratory symptoms/decreased lung function following bronchoscopy (Respiratory, thoracic and mediastinal disorders) | 6 (28) | 5 (84) | 5 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No